CLINICAL TRIAL: NCT07037407
Title: Accuracy Assessment of Intraoral Scan Versus Conventional Impression in Edentulous Patients With Flabby Ridges: A Prospective Clinical Study
Brief Title: Intraoral Scan Versus Conventional Impression in Edentulous Patients With Flabby Ridges
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Dina ElAwady, Associate Prof Of Prosthodontics, October University for Modern Sciences and Arts
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: MSA University REC-D4210-4
Record Dates: First submitted 2025-06-12; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Edentulism; Edentulous Alveolar Ridge; Edentulous Alveolar Ridge With Labial Resorption; Flabby Ridge
Keywords: Flabby ridge; IOS

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- WTI (Active Comparator): Control: Window technique for Maxillary flabby ridge using two consistencies of PVS impression material then poured to obtain a stone model which will be scanned using a laboratory extra oral scan to convert it into an STL file (WTI)
  Interventions: Procedure: WTI
- IOS (Experimental): intra oral scanning of flabby ridge
  Interventions: Procedure: IOS

INTERVENTIONS:
Procedure: IOS — Intra oral scanning
  Arms: IOS
Procedure: WTI — window technique Impression
  Arms: WTI

SUMMARY:
In vivo prospective clinical study will be designed, 12 participants will be included. After intraoral scanning, a conventional impression is made for each patient. The groups will be compared for accuracy.

DETAILED DESCRIPTION:
* Recruit 12 eligible edentulous patients
* Scanning Process: Perform five intraoral scans (IOS) of the maxillary flabby ridges for each patient.

  . WTI: perform five WTI for each patient
* STL Export: Export scans and corresponding cast scans obtained via the Window Technique Impression (WTI) as STL files using the intraoral scanner software.
* 3D Distance Measurement: Import IOS and cast STL files into Geomagic Wrap 2017 for a two-phase best-fit alignment, using the Cast scan as the reference for evaluating trueness and precision.
* Comparison of Scans:

  * Compare the IOS scan and corresponding cast scan obtained via the Window Technique Impression (WTI) to calculate trueness -compare WTI and corresponding cast scan obtained via the Window Technique Impression (WTI) to calculate trueness-
  * Compare each of the five IOS impressions by using each scan as a reference against the others to calculate precision.
  * Compare each of the five WTI impressions by using each scan as a reference against the others to calculate precision. • Deviation Analysis: Generate a color difference map of each superimposition for visual analysis of deviation patterns.

ELIGIBILITY:
Inclusion Criteria:Inclusion criteria for participant selection will be as follows: 1. completely edentulous patients with maxillary flabby ridge; 2. Absence of infectious diseases; 3. Systemic good health (ASA-1/ASA-2). .; 4. Age between 50 and 75 years; 5. Willingness to cooperate throughout the data collection process.

Exclusion Criteria:Exclusion criteria included: 1. Presence of any remaining teeth; 2. Inability to comprehend the study's objectives and procedures; 3. ridge defect or lesion; 4. Postoperative scarring on the ridge; 5. Limitations in mouth opening.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-10-18 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
accuracy evaluation | 1 month
  Accuracy Evaluation: The accuracy of the digital impressions versus conventional impression based on trueness and precision will be evaluated.
  - Trueness: Trueness is the degree of agreement between the digital impression and the reference scan. To assess trueness, we will measure the deviation between the reference and scanned files.
  Precision: Precision is a statistical measure that quantifies the level of similarity between repeated samples within the same group. In the context of this study, the IOS impression STL files will be compared to each other in a manner similar to the previous comparisons

CONTACTS AND LOCATIONS:
Locations (1):
- October University for Modern Sciences and Arts, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No